CLINICAL TRIAL: NCT00654797
Title: Clinical Process Improvement With A Bedside Computerized Insulin Therapy Protocol For Blood Glucose Control (eProtocol-insulin) in Adult And Pediatric Intensive Care Unit Patients-Second Phase (Phase-2): Distribution and Implementation of Validated eProtocol-insulin in Naïve ICUs
Brief Title: Improving Blood Glucose Control With a Computerized Decision Support Tool: Phase 2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01-HC-45210-2; HHSN268200425210C
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Critically Ill; Hyperglycemia
Keywords: Glucose; Insulin; computer; critical care
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eProtocol (Experimental)
  Interventions: Procedure: glucose control with computer generated recommendations

INTERVENTIONS:
Procedure: glucose control with computer generated recommendations — Insulin dosing will be recommended by the computer tools based on subject glucose values. Bedside clinicians will have the ablity to accept or reject the suggested dose.

SUMMARY:
The Purpose of this study is to:

1. Introduce the refined, validated, and safe computerized bedside decision support tool for blood glucose management in critically ill adult and pediatric ICU patients that was studied in Phase 1 into a second group of naïve ICUs, none of which participated in eProtocol-insulin development, refinement or validation
2. Monitor how often low blood sugar levels occur during use of the bedside tool.
3. Determine how the computerized tool effects the workload of the ICU nurses.

DETAILED DESCRIPTION:
In the current second phase of this project (Phase-2), we will introduce the refined, validated, and safe eProtocol-insulin into a second group of naïve ICUs, none of which participated in eProtocol-insulin development, refinement or validation. Our primary goal in this second phase is to determine the feasibility of exporting this tool to naïve ICU environments. In this second phase we will also compare the effects of the eProtocol-insulin and ordinary care approaches to glucose control on the bedside nurse's experience.

This second phase will be a prospective cohort study. We will determine the feasibility of distributing eProtocol-insulin and will further validate eProtocol-insulin in >4 adult and >4 pediatric ICUs. If necessary we will modify eProtocol-insulin with an iterative refinement process, with Institutional Review Board (IRB) and independent Data and Safety Monitoring Board (DSMB) oversight. eProtocol-insulin will be considered refined if >90% of the instructions are accepted and if the percent of glucose values between 70 and 110 mg/dl (3.9-6.1 mMol/L) are equivalent to our Phase-1 refinement and validation experience of 46%%, and if the rate of glucose values < 40 mg/dl (2.2 mMol/l) is less than 0.5% of glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric ICU: Proposed indications by pediatric clinicians at participating ICUs for glucose control in their ICUs would include patients who require mechanical ventilation for greater than 24 hours and/or require a vasoactive infusion (e.g. dopamine >3 mg/kg/min, dobutamine, epinephrine, or vasopressin).
2. Adult ICUs: Proposed indications by clinicians in participating ICUs for glucose control in participating adult ICUs include critically ill patients with an anticipated ICU length of stay of 3 or more days.

Exclusion Criteria:

1. Pregnancy (negative pregnancy test required for females of child-bearing age)
2. Age less than one month
3. Inborn errors of metabolism that the clinician suspects will affect glucose homeostasis
4. Acute or chronic liver disease with any documented episode of blood or plasma glucose <60 mg/dl within the 24 hours prior to study entry
5. Diabetic Ketoacidosis (critically ill patients with insulin dependent diabetes not in ketoacidosis will be eligible if attending physicians intend to use intravenous insulin as part of ordinary care)
6. Severe chronic liver disease (Child-Pugh score >10)

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable for feasibility during Phase-2 will be the acceptability of the eProtocol-insulin instructions (compliance of bedside clinicians with instructions). Proportion of glucose values < 40 mg/dl. | 1 year

SECONDARY OUTCOMES:
Proportion of glucose determinations between 70 and 110 mg/dl (3.9-6.1 mMol/L) (efficacy) | 1 year
Time to reach the 80-110 mg/dl target | 1 year
Nursing perception of workload in comparison to ordinary care (efficacy and feasibility) | 1 year
Proportion of glucose values 41-60 mg/dl | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Morris, MD, Principal Investigator — Intermountain Medical Center, Murray, Utah
Locations (10):
- United States (10):
  - Childrens Hospital Centeral California, Madera, California
  - Childrens Hospital of Minnesota - St. Paul, Saint Paul, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cornell University Medical College, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas